CLINICAL TRIAL: NCT00149266
Title: Randomized Controlled Trial to Evaluate Surgical Approaches to Gastric Cancer Invading the Esophagus (JCOG9502)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG9502; C000000122
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Gastric Neoplasm
Keywords: stomach neoplasms; lymph node resection; cardia; thoracotomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Surgery: abdominal and transhiatal approach
Procedure: Surgery: left thoraco-abdominal approach

SUMMARY:
To compare left thoraco-abdominal approach with abdominal and transhiatal approach to cardia or subcardia cancer

DETAILED DESCRIPTION:
For gastric cancers with esophageal invasion (Siewert type II and III), thoraco-abdominal approach has shown better survival results than abdominal approach in retrospective analyses. However, patients having mediastinal nodal metastasis have poor prognosis and the benefit of thoraco-abdominal approach is still controversial. We evaluated the two approaches in a prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

1. histologically proven adenocarcinoma
2. 75 years old or younger
3. forced expiratory volume in one second ≥ 50 %
4. arterial oxygen pressure in room air ≥ 70 mmHg
5. clinically T2/T3/T4 with ≤3 cm esophageal invasion
6. written consent

Exclusion Criteria:

1. Carcinoma in the remnant stomach
2. Borrmann type 4 (linitis plastica)
3. synchronous or metachronous malignancy in other organs except for cervical carcinoma in situ and colorectal focal cancer in adenoma
4. history of left thoracotomy, or left pleural adhesion
5. past history of myocardial infarction or positive results of exercise ECG
6. liver cirrhosis, or chronic liver disease with indocyanine green test ≥15%

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 1995-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
overall survival

SECONDARY OUTCOMES:
relapse-free survival
operative morbidity and mortality
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuru Sasako, MD, Study Chair — Gastric Surgery Division, National Cancer Center Hospital
Locations (1):
- National Cancer Center Hospital, 5-1-1 Tsukiji, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Result] Sasako M, Sano T, Yamamoto S, Sairenji M, Arai K, Kinoshita T, Nashimoto A, Hiratsuka M; Japan Clinical Oncology Group (JCOG9502). Left thoracoabdominal approach versus abdominal-transhiatal approach for gastric cancer of the cardia or subcardia: a randomised controlled trial. Lancet Oncol. 2006 Aug;7(8):644-51. doi: 10.1016/S1470-2045(06)70766-5. PMID 16887481
- [Derived] Kurokawa Y, Sasako M, Sano T, Yoshikawa T, Iwasaki Y, Nashimoto A, Ito S, Kurita A, Mizusawa J, Nakamura K; Japan Clinical Oncology Group (JCOG9502). Ten-year follow-up results of a randomized clinical trial comparing left thoracoabdominal and abdominal transhiatal approaches to total gastrectomy for adenocarcinoma of the oesophagogastric junction or gastric cardia. Br J Surg. 2015 Mar;102(4):341-8. doi: 10.1002/bjs.9764. Epub 2015 Jan 21. PMID 25605628
- [Derived] Kurokawa Y, Sasako M, Sano T, Shibata T, Ito S, Nashimoto A, Kurita A, Kinoshita T; Japan Clinical Oncology Group. Functional outcomes after extended surgery for gastric cancer. Br J Surg. 2011 Feb;98(2):239-45. doi: 10.1002/bjs.7297. PMID 21104822
- See also: Related Info — http://www.jcog.jp/